CLINICAL TRIAL: NCT06296056
Title: Single-center, Phase 1 Clinical Trial Evaluating the Safety and Preliminary Efficacy of a Combination Cellular Immunotherapy in Patients With Metastatic (Stage IV) Solid Tumors Refractory to standard-of Care Therapies.
Brief Title: Phase I Trial of Combined Immune Cell Therapy for Metastatic Stage IV Solid Tumors (SDH-Combi)
Acronym: SDH-Combi
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul Hospital (Other)
Responsible Party: Principal Investigator, Nyamdavaa Tuul, Director, Seoul Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDH-Combi; Mongolian IRB (Other: 24/094)
Record Dates: First submitted 2024-02-20; First posted 2024-03-06 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors; Metastatic
Keywords: immune cell therapy; dendritic cell; natural killer cell; cytotoxic T lymphocytes
MeSH Terms: conditions — Neoplasm Metastasis | interventions — beriplast P combi set

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SDH-Combi (Experimental): natural killer (NK) cells and cytotoxic T lymphocytes (CTLs)
  Interventions: Biological: Combi

INTERVENTIONS:
Biological: Combi — Biological immune cell therapy

SUMMARY:
To evaluate the safety and potential efficacy of combined immune cell therapy in patients with stage IV solid tumors who have failed standard treatment and have unresectable lesions or metastatic lesions.

DETAILED DESCRIPTION:
The combined immune cell therapy has a strong potential to improve treatment outcomes in several cancers, but problems related to manufacturing complexity, immunocompatibility, and poteintial toxicity may also arise. This clinical study was designed to address these challenges and to establish the safety and potential efficacy of combined immune cell therapy for unresectable solid tumors. This is a phase I study to evaluate the safety and potential efficacy of combined immune cell theapy, and obtain the recommended dose and infusion plan.

ELIGIBILITY:
Inclusion Criteria:

* Those who have been histologically or cytologically confirmed as adenocarcinoma among solid tumors
* Those with at least one measurable or evaliable lesion by RECIST v1.1
* Those who fail standard treatment for metastatic solid tumors (failure of treatment is defined as failure of not only progression of the disease or recurrence after treatment, but also unacceptable side effects or maintenance of the treatment process)
* ECOG performance status 0 or 1 person
* A person who can draw about 100 cc of whole blood for the manufacture of immune cells

  * Weight: More than 50 kg for men and more than 35 kg for women
  * Hb: 9.0 g/dL or higher (registerable if hemoglobin levels recover to 10.0 g/dL or higher during the screening period); however, transfusions within 7 days prior to screening to meet this standard are not allowed)
* Appropriate contraceptive regimen up to 2 months after clinical research drug administration
* A person who voluntarily decides to participate after receiving a sufficient explanation for this clinical study and agrees in writing

Exclusion Criteria:

* Brain Metastasis patients who have symptoms or need treatment [However, patients with stable brain metastasis who have no symptoms and do not need treatment (excluding anticonvulsants in maintenance therapy) can register]
* A person with a systemic disease that is inappropriate to administer anticancer drugs according to the researcher's judgment
* Those with the following cardio-cerebrovascular diseases as of the time of screening
* a person who is HIV-positive
* Those determined that the researcher was not suitable for participation in this clinical study as a result of the active infection (HBV, HCV) test
* a person with acute or severe infection
* Those who have autoimmune diseases or have a history of chronic or recurrent autoimmune diseases
* Those with a history of organ transplants
* a hematopoietic stem cell transplant patient

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-06-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) | 6 months
  All AEs will be collected and graded according to NCI-CTCAE v5.0. Data will be reported as the number and percentage of participants experiencing ≥1 AE.
Number of participants with serious adverse events (SAEs) | 6 months
  SAEs will be assessed for type, severity, and relationship to the investigational product. Reported as the number and percentage of participants experiencing ≥1 SAE.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) assessed by RECIST v1.1 | 6 months
  Defined as the proportion of participants with Complete Response (CR) or Partial Response (PR) according to RECIST v1.1. Reported as a percentage of evaluable participants.
Disease Control Rate (DCR) assessed by RECIST v1.1 | 6 months
  Defined as the proportion of participants achieving CR, PR, or Stable Disease (SD). Reported as a percentage of evaluable participants.
Change from baseline in EORTC QLQ-C30 global health status/quality of life score | 6 months
  Change from baseline to 6 months in the global health status/QoL domain of the EORTC QLQ-C30 questionnaire (0-100 scale; higher score indicates better outcome). Reported as mean change from baseline with standard deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Hospital, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: No